CLINICAL TRIAL: NCT00991679
Title: Expression of CXCL9, CXCL10, CXCL11, and CXCR3 in the Tear Film and Ocular Surface of Patients With Dry Eye Syndrome
Brief Title: CXCL9, CXCL10, CXCL11, and CXCR3 in Dry Eye Syndrome
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Kyung-Chul Yoon, MD/ Assisted professor, Department of Ophthalmology, Chonnam National University Medical School and Hospital, Gwangju, South Korea
Other Study IDs: I-2007-12-111
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye syndrome; CXCL9 chemokine; CXCL10 chemokine; CXCL11 chemokine; CXCR3 receptor
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tears, conjunctiva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal control subjects: Normal control subjects who did not show the clinical symptom and findings of dry eye syndrome.
- dry eye patients: Patients with dry eye syndrome who had symptoms of dry eye for more than 3 months, low tear film break up time (BUT, ≤7 sec), low Schirmer test (<10 mm), low tear clearance rate (<8X), and positive fluorescein or rose bengal vital staining (≥3) and were not treated with anti-inflammatory agents such as topical cyclosporine or steroids were included in the study.

SUMMARY:
The aim of this study is to investigate the expression of CXCL9, CXCL10, CXCL11, and CXCR3 in the tear film and ocular surface of patients with dry eye syndrome.

Thirty-three patients with dry eye (16 Sjögren's syndrome and 17 non-Sjögren's syndrome patients) and 15 control subjects were recruited. The concentrations of CXCL9, CXCL10, and CXCL11 in tears were measured using enzyme-linked immunosorbent assay. The correlation between chemokine levels and tear film and ocular surface parameters was analyzed. Expression of CXCL9, CXCL10, CXCL11, and CXCR3 in the conjunctiva was evaluated using immunohistochemistry. Flow cytometry was performed to count CXCR3+ cells and CXCR3+CD4+ cells in the conjunctiva.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of dry eye syndrome

Exclusion Criteria:

* active ocular infection or inflammation not associated with dry eye
* drug toxicity
* contact lens wear
* ocular allergy
* ocular surgery within the last 3 months
* lid or lash abnormalities

Ages: 24 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Chul Yoon, MD, PhD, Study Director — Department of Ophthalmology, Chonnam National University Medical School and Hospital, Gwangju, South Korea
Locations (1):
- Chonnam National University Hospital, Gwangju, Chonnam, South Korea

REFERENCES:
- [Result] Yoon KC, De Paiva CS, Qi H, Chen Z, Farley WJ, Li DQ, Pflugfelder SC. Expression of Th-1 chemokines and chemokine receptors on the ocular surface of C57BL/6 mice: effects of desiccating stress. Invest Ophthalmol Vis Sci. 2007 Jun;48(6):2561-9. doi: 10.1167/iovs.07-0002. PMID 17525185
- [Result] Wallace GR, John Curnow S, Wloka K, Salmon M, Murray PI. The role of chemokines and their receptors in ocular disease. Prog Retin Eye Res. 2004 Jul;23(4):435-48. doi: 10.1016/j.preteyeres.2004.04.004. PMID 15219876
- [Result] Pflugfelder SC, Jones D, Ji Z, Afonso A, Monroy D. Altered cytokine balance in the tear fluid and conjunctiva of patients with Sjogren's syndrome keratoconjunctivitis sicca. Curr Eye Res. 1999 Sep;19(3):201-11. doi: 10.1076/ceyr.19.3.201.5309. PMID 10487957
- [Derived] Yoon KC, Park CS, You IC, Choi HJ, Lee KH, Im SK, Park HY, Pflugfelder SC. Expression of CXCL9, -10, -11, and CXCR3 in the tear film and ocular surface of patients with dry eye syndrome. Invest Ophthalmol Vis Sci. 2010 Feb;51(2):643-50. doi: 10.1167/iovs.09-3425. Epub 2009 Oct 22. PMID 19850844